CLINICAL TRIAL: NCT06187038
Title: Effects of Including a Chronic Pain Neuroscience Education Program for Individuals With Knee OA: Randomized, Blinded Clinical Trial
Brief Title: Effects of Including a Chronic Pain Neuroscience Education Program for Individuals With Knee OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 70408123.1.0000.5511
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise group (Active Comparator): The therapeutic exercise program will include warm-up, resistance, neuromuscular, mobility, and balance exercises. Over ten weeks, two sessions of the therapeutic exercise program will be carried out individually, lasting approximately 60 minutes each-a total of 20 therapeutic exercise sessions. Therapeutic exercise sessions will be carried out at least 24 hours between sessions. The therapeutic exercises will be performed in up to three sets of 8-12 repetitions or 30-60 seconds each, with rest intervals of 90 seconds between sets.
  Interventions: Other: Therapeutic exercises
- Therapeutic exercise group and pain neuroscience education program (Experimental): The therapeutic exercise program will include warm-up, resistance, neuromuscular, mobility, and balance exercises. Over ten weeks, two sessions of the therapeutic exercise program will be carried out individually, lasting approximately 60 minutes each-a total of 20 therapeutic exercise sessions. Therapeutic exercise sessions will be carried out at least 24 hours between sessions. The therapeutic exercises will be performed in up to three sets of 8-12 repetitions or 30-60 seconds each, with rest intervals of 90 seconds between sets. The chronic pain neuroscience education program will be based on three domains. Making sense of pain, exposure with control, and lifestyle changes.
  Interventions: Other: Therapeutic exercises; Other: Therapeutic exercises + pain neuroscience education program

INTERVENTIONS:
Other: Therapeutic exercises — The therapeutic exercise program will include warm-up, resistance, neuromuscular, mobility, and balance exercises. Over ten weeks, two sessions of the therapeutic exercise program will be carried out individually, lasting approximately 60 minutes each-a total of 20 therapeutic exercise sessions. Therapeutic exercise sessions will be carried out at least 24 hours between sessions. Therapeutic exercises will be performed in up to three sets of 8-12 repetitions or 30-60 seconds each, with rest intervals of 90 seconds between sets.
Other: Therapeutic exercises + pain neuroscience education program — In addition to the therapeutic exercise protocol previously reported in the control group, research participants allocated to the experimental group will undergo an education program in the neurosciences of chronic pain carried out one day a week between the two therapeutic exercise sessions lasting ten weeks.
  The chronic pain neuroscience education program will be based on three domains. Making sense of pain, Exposure with control, and Lifestyle changes also urge modifications aimed at improving sleep, stress, and anxiety.
  Arms: Therapeutic exercise group and pain neuroscience education program

SUMMARY:
Research participants diagnosed with knee osteoarthritis will be randomized through a draw using sealed opaque envelopes indicating two groups: 1. therapeutic exercises, 2. therapeutic exercises + chronic pain neuroscience education program. The primary outcome will be functional performance using a patient-reported measure, the Knee Injury and Osteoarthritis Outcome Score (KOOS).

The selected secondary outcomes will be pain intensity by the numerical pain scale (END), physical function reported by the patient by the patient-specific functional scale (EFEP), Pain self-efficacy questionnaire (PSEQ), functional mobility by the timed up and test (TUG), general effect perceived through the global perception scale (EPG), muscle strength through Maximum Voluntary Isometric Contraction (MVIC) and functionality and disability through the World Health Organization Disability Assessment Schedule (WHODAS).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of knee osteoarthritis (knee pain for > 3 months
* Morning stiffness <30 minutes
* Crepitus
* Bone tenderness, and absence of palpable heat and/or diagnosis established radiographically (determined by Kellgren and Lawrence grade 1 to 3 on a scale 1 up to 4)

Exclusion Criteria:

* Hip OA
* severe osteoporosis
* Fibromyalgia
* Medical history of tumors or cancer
* Active inflammatory joint diseases (rheumatoid arthritis, gout)
* Undergoing any lower extremity joint replacement
* Neurological diseases (Parkinson's disease, stroke, Multiple Sclerosis, muscular dystrophy, motor neuron disease, Alzheimer's disease, cognitive and cardiopulmonary impairment that may prevent or limit the performance of exercises, use of a gait assistance device, history of recent knee trauma.
* Having undergone any form of treatment involving physiotherapy, intra-articular corticosteroids, anti-inflammatories or chondroprotective in the last six months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional disability | Change from Baseline, after 10 weeks of intervention and 4 weeks after the end of the intervention.
  Knee Injury and Osteoarthritis Outcome Score (KOOS). It aims to evaluate the domains of pain, symptoms, activities of daily living, function related to recreation and sports, and quality of life related to the knee. Totaling 42 items, each item must be answered using a Likert scale that ranges from 0 (best score) to 4 (worst score), and the score for each subscale ranges from 0 (worst score) to 100 (best score).

SECONDARY OUTCOMES:
Numerical Pain Scale | Change from Baseline, after 10 weeks of intervention and 4 weeks after the end of the intervention.
  The Numerical rating pain scale, a simple, easily administered scale evaluates the perceived intensity of pain, using an 11-point scale from 0, representing 'no pain', to 10, which is the 'worst possible pain'.
Functional self-perception | Change from Baseline, after 10 weeks of intervention and 4 weeks after the end of the intervention.
  Pain self-efficacy questionnaire, structured into 10 items where each item is evaluated by selecting a number on a 7-point numerical scale (scores from 0 to 6), where 0 means "not at all confident" and 6 means "completely confident". The items cover different functions, from work, social activities, domestic tasks and coping with pain without medication. A total score is calculated from the sum of the scores for each of the 10 items, producing a total score that ranges from 0 to 60. Higher scores reflect stronger self-efficacy beliefs.
Self-perceived functionality | Change from Baseline, after 10 weeks of intervention and 4 weeks after the end of the intervention.
  Patient Specific Functional Scale. An easy-to-apply self-report instrument, validated for measuring disability related to specific tasks identified by the individual. The scale is made up of 11 (eleven) numbers, graduated from 0 (zero) to 10 (ten), where 0 (zero) represents inability to perform the activity and ten (ten) the ability to perform the activity at the level prior to the current condition.
Maximum voluntary isometric contraction | Change from Baseline, after 10 weeks of intervention and 4 weeks after the end of the intervention.
  manual dynamometer portable (Lafayette Manual Muscle System, Modelo 01165, Lafayette Instrument Company, Lafayette, IN). Four 5-second readings will be taken during maximal voluntary isometric contraction (MVIC) with a 30-second rest period between contractions. The first CIVM will familiarize the volunteer with carrying out the task. A new set of readings will be taken if a volunteer can perform three contractions with at least 10% variability. Strong and constant verbal stimuli will be used throughout the test. Always with the research participants' hands positioned crossed on the chest. Thus, bilateral assessments of the muscles, quadriceps, and gluteus medius will be carried out. The order of CIVM readings will be randomized to avoid collection bias. The research participant will remain in lateral decubitus with a pillow positioned between the legs, with the limb to be tested superiorly in a neutral position.
Dynamic balance | Change from Baseline, after 10 weeks of intervention and 4 weeks after the end of the intervention.
  Iimed up and go test, research participants will be instructed to get up from a chair, walk 3 meters comfortably and safely, come back and sit down in the chair. The time taken to complete this task will be measured using a stopwatch that will be started after the verbal command 'go' and stopped when the participant returns to the initial sitting position. A first attempt will be made to familiarize the participant with the procedure. Two assessments will then be carried out. The average of the two assessments will be recorded for later data analysis.
Global Perception of Change scale | Change from Baseline, after 10 weeks of intervention and 4 weeks after the end of the intervention.
  The perception of the global effect of the treatment by the research participant will be evaluated by the Global Perception of Change scale. The Global Perception of Change scale is a direct scale on the patient's self-perception when the intervention is performed. This scale consists of 11 points, ranging from -5 (worsening compared to the start of treatment), 0 (neutral) and +5 (improvement compared to the start of treatment), using the Portuguese version.
Functionality | Change from Baseline, after 10 weeks of intervention and 4 weeks after the end of the intervention.
  The WHODAS 2.0 short version (12 items) is a generic self-report assessment instrument developed by the World Health Organization (WHO) to assess functionality and disability during the last 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Cid Gomes, PhD, Principal Investigator — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Make data available remotely in digital cloud storage.